CLINICAL TRIAL: NCT00363051
Title: An Open Label, Stratified, Single-arm Phase II Study of Everolimus in Patients With Advanced Pancreatic Neuroendocrine Tumor (NET) After Failure of Cytotoxic Chemotherapy
Brief Title: Safety/Efficacy of Everolimus in Adults With Advanced Pancreatic Neuroendocrine Cancer Not Responsive to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2239
Record Dates: First submitted 2006-08-02; First posted 2006-08-15 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Islet Cell Carcinoma; Neuroendocrine Carcinoma; Neuroendocrine Tumor; Pancreatic Neoplasms
Keywords: Pancreatic; Tumor; Islet Cell; Carcinoma; Neuroendocrine; Endocrine; Atypical Carcinoid; RADIANT1; RADIANT-1
MeSH Terms: conditions — Carcinoma, Islet Cell; Carcinoma, Neuroendocrine; Neuroendocrine Tumors; Pancreatic Neoplasms; Neoplasms; Carcinoma | interventions — Everolimus

ARMS (1):
- Everolimus 10 mg (Experimental): Stratum 1 patients who were not receiving regular Octreotide Depot therapy. These patients were to receive everolimus monotherapy at 10 mg/day.
  Stratum 2 patients who were to receive everolimus 10 mg/day in addition to continuing their entry dose of Octreotide Depot therapy.
  Patients were instructed to take two 5 mg tablets of everolimus orally with a glass of water, once daily (preferably in the morning). Dosing was strongly recommended to occur at the same time every day.
  Interventions: Drug: Everolimus 10 mg; Drug: Octreotide Depot

INTERVENTIONS:
Drug: Everolimus 10 mg — Participants took two 5 mg tablets of Everolimus orally with a glass of water, once daily (preferably in the morning) in a fasting state or after no more than a light, fat-free meal. Dosing was to occur at the same time each day. If vomiting occurred, the vomited dose was not to be replaced.
  Other Names: RAD001
Drug: Octreotide Depot

SUMMARY:
The purpose of this study was to assess the efficacy and safety of everolimus in the treatment of advanced pancreatic neuroendocrine tumor (NET) not responsive to cytotoxic chemotherapy. All patients were treated with everolimus until either tumor progression was documented using a standard criteria that measures tumor size called Response Evaluation Criteria in Solid tumors (RECIST), or until unacceptable toxicity occurred, or until the patient or investigator requested discontinuation of treatment.

DETAILED DESCRIPTION:
This was a stratified two-stage, single-arm, phase 2 study of treatment with everolimus in patients with advanced (unresectable or metastatic) pancreatic neuroendocrine tumor (NET) after failure of cytotoxic chemotherapy.

Stratum 1, consisted of patients not receiving chronic Octreotide Depot therapy, will receive everolimus monotherapy at 10 mg/day.

Stratum 2, consisting of patients with tumors that have progressed during Octreotide Depot treatment will continue their entry dose of Octreotide Depot plus everolimus 10 mg/day.

ELIGIBILITY:
Inclusion criteria for both strata:

* Advanced (unresectable or metastatic) biopsy-proven pancreatic Neuroendocrine tumor (NET)
* Confirmed low-grade or intermediate-grade neuroendocrine carcinoma
* Objective disease progression by Response Evaluation Criteria in Solid tumors (RECIST) criteria while receiving cytotoxic chemotherapy or at any time after receiving an adequate course of cytotoxic chemotherapy (i.e., at least 3 consecutive cycles or months of treatment with the same cytotoxic drug or regimen)
* Presence of at least one measurable disease using RECIST criteria at screening (computer tomography [CT] or Magnetic resonance imaging [MRI])
* Adequate bone marrow, liver and kidney function
* WHO Performance Status 0-2.

Inclusion criteria for Stratum 2 only:

* Meet all inclusion criteria defined above for both strata.
* Receiving treatment (at least 3 consecutive months) with Octreotide Depot.
* In addition to documentation of progressive disease on or after chemotherapy, patients in stratum 2 must have documented objective progression of disease while receiving Octreotide Depot.

Exclusion criteria for both strata:

* Anticancer therapy within 3 weeks of enrollment.
* Patients with poorly differentiated neuroendocrine carcinoma
* Hepatic artery embolization within the last 6 months
* Prior therapy with everolimus or other rapamycins (sirolimus, temsirolimus)
* Other concurrent malignancy
* Other serious intercurrent infections or nonmalignant uncontrolled medical illnesses

Exclusion Criterion for Stratum 1 only:

• Received treatment with Octreotide Depot or any other long-acting somatostatin analogue in the 60 days prior to enrollment or any short-acting somatostatin analogue in the two weeks prior to enrollment.

Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (54):
- United States (20):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - USC Medical Center, Los Angeles, California
  - Cedars-Sinai Outpatient Cancer Center/Samuel Oschin Comprehensive Cancer Inst., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University of Miami, Miami, Florida
  - H. Lee Moffit Cancer Center & Research Institute, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - LSUHC Multispecialty Clinic, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Lynn Ratner, M.D., New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Arthur G. James Cancer Hospital/Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - M. D Anderson Cancer Center, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Santa Fe
- Australia (3):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Herston
  - Novartis Investigative Site, Kogarah
- Novartis Investigative Site, Leuven, Belgium
- Canada (5):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (6):
  - Novartis Investigative Site, Billancourt
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Ulm
- Italy (5):
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Modena
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Rome
  - Novartis Investigative Site, Torrette Di Ancona
- Novartis Investigative Site, Gronigen, Netherlands
- Spain (3):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Uppsala, Sweden

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/webapp/etrials/searchTrial.do?t=i&trialID=525&diseaseID=92

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1: Everolimus 10 mg: Stratum 1 patients who were not receiving regular Octreotide Depot therapy. These patients were to receive everolimus monotherapy at 10 mg/day. Patients were instructed to take two 5 mg tablets of everolimus orally with a glass of water, once daily (preferably in the morning). Dosing was strongly recommended to occur at the same time every day.
- Stratum 2: Everolimus 10 mg + Octreotide Depot: Stratum 2 participants who had received at least three consecutive months of Octreotide Long Acting Depot therapy prior to enrollment. These patients also received Everolimus 10 mg/day in addition to continuing their entry dose of Octreotide Depot.
  Patients were instructed to take two 5 mg tablets of everolimus orally with a glass of water, once daily (preferably in the morning). Dosing was strongly recommended to occur at the same time every day.
Period: Overall Study
Arm/Group | Stratum 1: Everolimus 10 mg | Stratum 2: Everolimus 10 mg + Octreotide Depot
Started | 115 | 45
Completed | 77 (Patients with documented disease progression per RECIST criteria) | 23
Not Completed | 38 | 22
Not completed — Adminstrative problems | 1 | 1
Not completed — Adverse Event | 21 | 12
Not completed — New Cancer Therapy | 2 | 1
Not completed — Withdrawal by Subject | 11 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Stratum 2: Everolimus 10 mg + Octreotide Depot: Stratum 2 participants who had received at least three consecutive months of Octreotide Long Acting Depot therapy prior to enrollment. These patients also received Everolimus 10 mg/day in addition to continuing their entry dose of Octreotide Depot.
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Everolimus 10 mg | Stratum 2: Everolimus 10 mg + Octreotide Depot | Total
Number analyzed (Participants) | 115 | 45 | 160
Age Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.8) | 53.64 (12.478) | 54.33 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 21 | 70
  Male | 66 | 24 | 90

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate: Percentage of Participants With Best Over All Response of Complete Response or Partial Response by Central Radiology Review (Stratum 1) Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response rate was defined by RECIST criteria: Partial response (PR) must have ≥ 30% decrease in the sum of longest diameter of all target lesions, from the baseline sum. Complete response (CR) must have disappearance of all target and non-target lesions. For CR or PR, tumor measurements must be confirmed by 2nd assessments within 4 weeks. Progression = 20% increase in the sum of longest diameter of all target lesions, from smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions.
Time Frame: from date of randomization/start of treatment until first documented response confirmed 4 weeks later( at least 3 months)
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1: Everolimus 10 mg
Number analyzed (Participants) | 115
percentage of participants | 9.6 [4.9 to 16.5]

2. Secondary Outcome: Duration of Overall Response (Stratum 1) Based on Response Evaluation Criteria in Solid Tumors (RECIST)- Central Radiology Review
Description: Duration of overall response applies only to patients whose best overall response was complete response (CR) or partial response (PR):
  * Complete Response (CR) = at least two determinations of CR at least 4 weeks apart before progression.
  * Partial response (PR) = at least two determinations of PR or better at least 4 weeks apart before progression.
  Progression = 20% increase in the sum of the longest diameter of all target lesions, from the smallest sum of longest diameter of all target lesions recorded at or after baseline; or a new lesion; or progression of non-target lesions
Time Frame: from date of first documented confirmed response to time to progression, at least 3 months
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of everolimus. Only those patients whose best overall response was complete response (CR) or partial response (PR) were included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 1: Everolimus 10 mg
Number analyzed (Participants) | 11
Months | 10.64 [9.79 to NA] — The upper limit was not estimable in the study as it is longer than duration of study.

3. Secondary Outcome: Duration of Overall Response (Stratum 2) Based on Response Evaluation Criteria in Solid Tumors (RECIST)- Central Radiology Review
Description: as for outcome 2
Time Frame: from date of first documented confirmed response to time to progression, at least 3 months
Population: Very low number of patients demonstrated a partial response, the median duration of response as per central review has not been calculated.
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 0

4. Secondary Outcome: Objective Response Rate: Percentage of Participants With Best Over All Response of Complete Response or Partial Response by Central Radiology Review (Stratum 2) Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: as for outcome 1
Time Frame: from date of randomization/start of treatment until first documented response confirmed 4 weeks later (at least 3 months)
Population: Full Analysis Set (FAS) was consisted of all patients who received at least one dose of everolimus.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 45
percentage of participants | 4.4 [0.5 to 15.1]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs), Death, Serious Adverse Events (SAEs)[Stratum 1]
Description: Adverse events are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: on or after the day of the first intake of study treatment to starting no later than 28 days after study treatment discontinuation, at least every month
Population: The safety population consists of all patients who received at least one dose of everolimus and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Stratum 1: Everolimus 10 mg
Number analyzed (Participants) | 115
Participants
  Adverse Events | 115
  Death | 10
  Serious Adverse Events | 63

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Death, Serious Adverse Events (SAEs) [Stratum 2]
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 45
Participants
  Adverse Events | 45
  Death | 2
  Serious Adverse Events | 27

7. Secondary Outcome: Time to Progression Free Survival (PFS) Per Central Radiology Review (Stratum 1)
Description: Progression free survival (PFS) is defined as the time from randomization to the date of first documented disease progression or death from any cause. The Kaplan-Meier estimate of the PFS survival function was constructed.
  Median PFS was obtained and displayed along with 95% confidence intervals.
Time Frame: from randomisation to dates of disease progression, death from any cause or last tumor assessment, reported between day of first patient randomised, 26 June 2006, until cut-off date 13 September 2010
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 1: Everolimus 10 mg
Number analyzed (Participants) | 115
Months | 9.69 [8.25 to 13.31]

8. Secondary Outcome: Time to Progression Free Survival (PFS) Per Central Radiology Review (Stratum 2)
Description: as for outcome 7
Time Frame: as for outcome 7
Population: The full analysis set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 45
Months | 16.69 [11.07 to NA] — The upper limit was not estimable in the study as it is longer than duration of study.

9. Secondary Outcome: Time to Overall Survival (OS)(Stratum 1)
Description: Overall survival measures the time of survival , with any response or disease progression, until death. The OS is defined as the time from date of start of treatment to date of death due to any cause.
  If a patient is not known to have died, survival was censored at the date of last contact. In each treatment stratum, the Kaplan-Meier estimate of the overall survival function was constructed.
Time Frame: from randomisation to dates of disease progression, death from any cause, reported between day of first patient randomised, 26 June 2006, until cut-off date 13 April 2012
Population: The full analysis set consisted of all patients who received at least one dose of everolimus.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 1: Everolimus 10 mg
Number analyzed (Participants) | 115
months | 28.78 [20.24 to 36.37]

10. Secondary Outcome: Time to Overall Survival (OS) (Stratum 2)
Description: as for outcome 9
Time Frame: as for outcome 9
Population: The full analysis set consisted of all patients who received at least one dose of everolimus.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 45
months | 38.77 [29.08 to NA] — The upper limit was not estimable in the study as it is longer than duration of study.

11. Secondary Outcome: Everolimus Trough Level Determination by Pharmacokinetics Parameter in Both Strata (Stratum 1 and 2)
Description: For all patients in both strata, a blood sample for everolimus trough level determination will be collected immediately prior to the everolimus administration on Cycle 1 Day 15, Cycle 2 Day 1, and every month thereafter. A treatment cycle was defined as 28 days of consecutive daily treatment with everolimus and treatment continued until tumor progression. It is critical that patients not take their daily everolimus dose before the sample is drawn.
Time Frame: Cycle 1 Day 15
Population: Full Analysis Set (FAS) is consisted of all patients who received at least one dose of everolimus. Patients with everolimus pharmacokinteic samples, with nonzero concentration, at Cycle 1 Day 15 were included
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Stratum 1: Everolimus 10 mg | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 92 | 30
ng/ml | 15.7 (15.82) | 17.3 (18.08)

12. Secondary Outcome: Effect of Octreotide Depot on the Trough Concentrations of Everolimus
Description: The effect of Octreotide Depot on the trough concentrations of everolimus was assessed at Cycle 1 Day 15.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1
Population: Full Analysis Set (FAS) is consisted of all patients who received at least one dose of everolimus. Patients with Octreotide Depot pharmacokinetic samples, with nonzero concentration, at Cycle 1 Day 1 or Cycle 2 Day 1 were included.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Stratum 2: Everolimus 10 mg + Octreotide Depot
Number analyzed (Participants) | 38
ng/ml
  Cycle 1 Day 1 (pre-treatment baseline) (n=37) | 3.2 (2.81)
  Cycle 2 Day 1 (n= 38) | 3.7 (3.47)

ADVERSE EVENTS:
Arm/Group | Stratum 1: Everolimus 10 mg | Stratum 2: Everolimus 10 mg + Octreotide Depot
Serious Adverse Events (participants affected / at risk) | 63/115 | 27/45
Other Adverse Events (participants affected / at risk) | 115/115 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Everolimus 10 mg (N=115) | Stratum 2: Everolimus 10 mg + Octreotide Depot (N=45)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Subileus (Gastrointestinal disorders) | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Asthenia (General disorders) | 6 | 0
Device dislocation (General disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 0
General physical health deterioration (General disorders) | 2 | 0
Hyperthermia (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 2
Performance status decreased (General disorders) | 2 | 0
Pyrexia (General disorders) | 6 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Serratia infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1
Ammonia increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Coma hepatic (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 3
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Everolimus 10 mg (N=115) | Stratum 2: Everolimus 10 mg + Octreotide Depot (N=45)
Anaemia (Blood and lymphatic system disorders) | 22 | 11
Leukopenia (Blood and lymphatic system disorders) | 10 | 2
Lymphopenia (Blood and lymphatic system disorders) | 10 | 0
Neutropenia (Blood and lymphatic system disorders) | 10 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 6
Conjunctivitis (Eye disorders) | 4 | 4
Vision blurred (Eye disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 38 | 9
Abdominal pain upper (Gastrointestinal disorders) | 25 | 7
Aphthous stomatitis (Gastrointestinal disorders) | 24 | 6
Ascites (Gastrointestinal disorders) | 9 | 0
Constipation (Gastrointestinal disorders) | 30 | 8
Diarrhoea (Gastrointestinal disorders) | 63 | 25
Dry mouth (Gastrointestinal disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 1
Flatulence (Gastrointestinal disorders) | 6 | 4
Haemorrhoids (Gastrointestinal disorders) | 2 | 3
Mouth ulceration (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 54 | 22
Steatorrhoea (Gastrointestinal disorders) | 1 | 3
Stomatitis (Gastrointestinal disorders) | 57 | 24
Toothache (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 40 | 12
Asthenia (General disorders) | 38 | 9
Chills (General disorders) | 10 | 4
Fatigue (General disorders) | 53 | 20
Non-cardiac chest pain (General disorders) | 6 | 1
Oedema peripheral (General disorders) | 34 | 14
Pain (General disorders) | 7 | 3
Pyrexia (General disorders) | 41 | 14
Bronchitis (Infections and infestations) | 4 | 4
Influenza (Infections and infestations) | 7 | 4
Nasopharyngitis (Infections and infestations) | 18 | 5
Pneumonia (Infections and infestations) | 4 | 3
Rhinitis (Infections and infestations) | 7 | 2
Sinusitis (Infections and infestations) | 12 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 4
Urinary tract infection (Infections and infestations) | 11 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 4
Alanine aminotransferase increased (Investigations) | 7 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 0
Blood alkaline phosphatase increased (Investigations) | 9 | 1
Blood creatinine increased (Investigations) | 1 | 6
Haemoglobin decreased (Investigations) | 4 | 3
International normalised ratio increased (Investigations) | 1 | 3
Weight decreased (Investigations) | 32 | 12
Decreased appetite (Metabolism and nutrition disorders) | 27 | 10
Dehydration (Metabolism and nutrition disorders) | 5 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 11 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 21 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Dizziness (Nervous system disorders) | 5 | 7
Dysgeusia (Nervous system disorders) | 14 | 7
Headache (Nervous system disorders) | 40 | 9
Anxiety (Psychiatric disorders) | 8 | 3
Confusional state (Psychiatric disorders) | 6 | 2
Depression (Psychiatric disorders) | 10 | 2
Insomnia (Psychiatric disorders) | 15 | 5
Nocturia (Renal and urinary disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Acne (Skin and subcutaneous tissue disorders) | 7 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 7
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 7
Rash (Skin and subcutaneous tissue disorders) | 54 | 21
Hypertension (Vascular disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis's agreements with it's investigators vary. However, Novartis does not prohibit any investigator from publishing. Any publication from a single-center site is postponed until the publication of the pooled data ( i.e. data from all sites) in the clinical trial.